CLINICAL TRIAL: NCT05012293
Title: Cognitive Fatigue, Self-Regulation, and Academic Performance: A Physiological Study
Acronym: FRAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: National Research Foundation, Singapore (Other Government); Ministry of National Development, Singapore (Other Government); Housing and Development Board, Singapore (Other Government)
Responsible Party: Principal Investigator, Georgios CHRISTOPOULOS, Associate Professor, Nanyang Technological University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COT-V4-2020-1-S003
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Fatigue; Mental Fatigue; Behavioral Performance; Heart Rate Variability; Skin Conductance; Academic Performance; Self-regulation
MeSH Terms: conditions — Mental Fatigue; Self-Control | interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Fatigue Manipulation (Experimental)
  Interventions: Other: Baseline; Other: Fatigue Manipulation

INTERVENTIONS:
Other: Baseline — 5-min urban park video clip (Presented on a TV)
Other: Fatigue Manipulation — 20-min 2-back task (Presented on a computer)

SUMMARY:
This study aims to examine the relationship among cognitive fatigue, self-regulation, and academic performance.

DETAILED DESCRIPTION:
1) Sievertsen et al. (2016) have demonstrated that standardised test performance decreased with every hour later in the day and increased after a break. Hence, we hypothesise that standardised test performance would vary as a function of physiological response during cognitive fatigue. 2) Martin et al. (2019) found that those who participate in more self-regulatory activity were less susceptible to the effects of cognitive fatigue. Hence, we hypothesise that greater self-regulation may moderate the relationship between cognitive fatigue and standardised test performance. Individual differences (i.e., age, gender, caffeine and food intake, body mass index, skin temperature, sleep quality, depression, anxiety, stress, baseline physiology and behavioural performance) will be examined and accounted for.

ELIGIBILITY:
Inclusion Criteria:

* Singapore-based
* Non-clinical
* 18-35years

Exclusion Criteria:

* Individuals with hearing difficulties or failing to meet the minimal threshold for normal hearing
* Individuals with a history of ear, developmental, neurological, or psychiatric disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 162 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
2-Back Task (Change) | during fatigue manipulation procedure
  Change in Accuracy over time
2-Back Task (Change) | during fatigue manipulation procedure
  Change in Reaction Time over time
Fatigue State Questionnaire | up to 5 mins after fatigue manipulation
  Fatigue State Questionnaire Score
Electrocardiograph (Change) | during fatigue manipulation procedure
  Change in Heart Rate Variability over time
Electrodermal Activity (Change) | during fatigue manipulation procedure
  Change in Skin Conductance Level over time
Electrodermal Activity (Change) | during fatigue manipulation procedure
  Change in Skin Conductance Response over time
Short Self-Regulation Questionnaire | up to 1 hour before fatigue manipulation
  Short Self-Regulation Questionnaire Score
Academic Performance | up to 1 hour before fatigue manipulation
  Self-reported Academic Results

CONTACTS AND LOCATIONS:
Locations (1):
- Cultural Science Innovations, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin K, Thompson KG, Keegan R, Rattray B. Are Individuals Who Engage in More Frequent Self-Regulation Less Susceptible to Mental Fatigue? J Sport Exerc Psychol. 2019 Oct 1;41(5):289-297. doi: 10.1123/jsep.2018-0222. PMID 31509795
- [Background] Sievertsen HH, Gino F, Piovesan M. Cognitive fatigue influences students' performance on standardized tests. Proc Natl Acad Sci U S A. 2016 Mar 8;113(10):2621-4. doi: 10.1073/pnas.1516947113. Epub 2016 Feb 16. PMID 26884183